CLINICAL TRIAL: NCT00113763
Title: An Open-label, Randomized, Phase 3 Clinical Trial of ABX-EGF Plus Best Supportive Care Versus Best Supportive Care in Subjects With Metastatic Colorectal Cancer
Brief Title: Evaluating Panitumumab (ABX-EGF) Plus Best Supportive Care Versus Best Supportive Care in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020408
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer; Metastases
Keywords: Metastatic Colorectal Cancer, Colon; Colorectal, Rectal Cancer, Cancer; Metastatic, EGFr, Clinical Trial; Panitumumab, ABX-EGF; Immunex, Abgenix, Amgen
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms; Neoplasms | interventions — Panitumumab

ARMS (2):
- Panitumumab plus best supportive care (Experimental): Panitumumab will be administered by intravenous infusion at a dose of 6 mg/kg once every 2 weeks until participants develop progressive disease or are unable to tolerate study drug. Participants will also receive best supportive care (BSC) as judged appropriate by the investigator and according to institutional guidelines.
  Interventions: Drug: Panitumumab
- Best Supportive Care (Other): Best supportive care will be defined in this study as the best care available as judged appropriate by the investigator and according to institutional guidelines and will include antibiotics, analgesics, radiation therapy for pain control (limited to bone metastases), corticosteroids, transfusions, psychotherapy, growth factors, palliative surgery, or any symptomatic therapy as clinically indicated. For the purpose of this study, best supportive care will not include anti-neoplastic chemotherapy.
  Interventions: Other: Best supportive care

INTERVENTIONS:
Other: Best supportive care — Best supportive care as site routine excluding: antineoplastic chemotherapy, investigational agents, anti-EGFr(Epidermal growth factor receptor) targeting agents other than ABX-EGF(Panitumumab), experimental or approved anti-tumor therapies (e.g. Avastin), chemotherapy, radiotherapy (with the exception of radiotherapy for pain control limited to bone metastases).
  Arms: Best Supportive Care
Drug: Panitumumab — Intravenous infusion at a dose of 6 mg/kg once every 2 weeks.
  Other Names: ABX-EGF
  Arms: Panitumumab plus best supportive care

SUMMARY:
The purpose of this study is to determine that panitumumab, using the proposed regimen, will safely increase progression free survival in patients with metastatic colorectal cancer who have failed available treatment options (i.e., patients who developed progressive disease or relapsed while on or after prior fluoropyrimidine, irinotecan and oxaliplatin chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of colorectal adenocarcinoma (diagnostic tissue obtained by tissue biopsy)
* Metastatic colorectal carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Documented evidence of disease progression during, or following treatment, with fluoropyrimidine, irinotecan and oxaliplatin chemotherapy for metastatic colorectal cancer
* Radiographic documentation of disease progression during or within 6 months following the most recent chemotherapy regimen
* Unidimensionally measurable disease
* Tumor expressing epidermal growth factor receptor (EGFr) by immunohistochemistry
* At least 2 but not more than 3 prior chemotherapy regimens for colorectal cancer
* Adequate hematologic, renal and hepatic function

Exclusion Criteria:

* Symptomatic brain metastases requiring treatment
* History or evidence of interstitial pneumonitis or pulmonary fibrosis
* Use of systemic chemotherapy or radiotherapy within 30 days prior to enrollment
* Prior epidermal growth factor receptor (EGFr) targeting therapies
* Prior anti-tumor therapies including prior experimental agents or approved anti-tumor small molecules and biologics of short (less than a week) serum half life within 30 days before enrollment, or prior experimental or approved proteins within 3 months before enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2009-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Bai JP, Bell R, Buckman S, Burckart GJ, Eichler HG, Fang KC, Goodsaid FM, Jusko WJ, Lesko LL, Meibohm B, Patterson SD, Puig O, Smerage JB, Snider BJ, Wagner JA, Wang J, Walton MK, Weiner R. Translational biomarkers: from preclinical to clinical a report of 2009 AAPS/ACCP Biomarker Workshop. AAPS J. 2011 Jun;13(2):274-83. doi: 10.1208/s12248-011-9265-x. Epub 2011 Mar 30. PMID 21448748
- [Background] Odom D, Barber B, Bennett L, Peeters M, Zhao Z, Kaye J, Wolf M, Wiezorek J. Health-related quality of life and colorectal cancer-specific symptoms in patients with chemotherapy-refractory metastatic disease treated with panitumumab. Int J Colorectal Dis. 2011 Feb;26(2):173-81. doi: 10.1007/s00384-010-1112-5. Epub 2010 Dec 29. PMID 21190026
- [Background] Peeters M, Siena S, Van Cutsem E, Sobrero A, Hendlisz A, Cascinu S, Kalofonos H, Devercelli G, Wolf M, Amado RG. Association of progression-free survival, overall survival, and patient-reported outcomes by skin toxicity and KRAS status in patients receiving panitumumab monotherapy. Cancer. 2009 Apr 1;115(7):1544-54. doi: 10.1002/cncr.24088. PMID 19189371
- [Background] Siena S, Peeters M, Van Cutsem E, Humblet Y, Conte P, Bajetta E, Comandini D, Bodoky G, Van Hazel G, Salek T, Wolf M, Devercelli G, Woolley M, Amado RG. Association of progression-free survival with patient-reported outcomes and survival: results from a randomised phase 3 trial of panitumumab. Br J Cancer. 2007 Dec 3;97(11):1469-74. doi: 10.1038/sj.bjc.6604053. Epub 2007 Nov 27. PMID 18040272
- [Background] Van Cutsem E, Peeters M, Siena S, Humblet Y, Hendlisz A, Neyns B, Canon JL, Van Laethem JL, Maurel J, Richardson G, Wolf M, Amado RG. Open-label phase III trial of panitumumab plus best supportive care compared with best supportive care alone in patients with chemotherapy-refractory metastatic colorectal cancer. J Clin Oncol. 2007 May 1;25(13):1658-64. doi: 10.1200/JCO.2006.08.1620. PMID 17470858
- [Derived] Safari M, Esmaeili H, Mahjub H, Roshanaei G. Estimation of treatment effect in presence of noncompliance and competing risks: a simulation study. Sci Rep. 2023 Aug 18;13(1):13477. doi: 10.1038/s41598-023-40538-2. PMID 37596461
- [Derived] Liao MZ, Prenen H, Dutta S, Upreti VV. The impact of hepatic and renal function on panitumumab exposures in patients with metastatic RAS wild-type colorectal cancer. Cancer Chemother Pharmacol. 2021 Oct;88(4):665-672. doi: 10.1007/s00280-021-04319-w. Epub 2021 Jul 2. PMID 34213592
- [Derived] Boeckx N, Koukakis R, Op de Beeck K, Rolfo C, Van Camp G, Siena S, Tabernero J, Douillard JY, Andre T, Peeters M. Effect of Primary Tumor Location on Second- or Later-line Treatment Outcomes in Patients With RAS Wild-type Metastatic Colorectal Cancer and All Treatment Lines in Patients With RAS Mutations in Four Randomized Panitumumab Studies. Clin Colorectal Cancer. 2018 Sep;17(3):170-178.e3. doi: 10.1016/j.clcc.2018.03.005. Epub 2018 Mar 8. PMID 29627309
- [Derived] Peeters M, Kafatos G, Taylor A, Gastanaga VM, Oliner KS, Hechmati G, Terwey JH, van Krieken JH. Prevalence of RAS mutations and individual variation patterns among patients with metastatic colorectal cancer: A pooled analysis of randomised controlled trials. Eur J Cancer. 2015 Sep;51(13):1704-13. doi: 10.1016/j.ejca.2015.05.017. Epub 2015 Jun 3. PMID 26049686
- [Derived] Poulin-Costello M, Azoulay L, Van Cutsem E, Peeters M, Siena S, Wolf M. An analysis of the treatment effect of panitumumab on overall survival from a phase 3, randomized, controlled, multicenter trial (20020408) in patients with chemotherapy refractory metastatic colorectal cancer. Target Oncol. 2013 Jun;8(2):127-36. doi: 10.1007/s11523-013-0271-z. Epub 2013 Apr 27. PMID 23625191
- [Derived] Amado RG, Wolf M, Peeters M, Van Cutsem E, Siena S, Freeman DJ, Juan T, Sikorski R, Suggs S, Radinsky R, Patterson SD, Chang DD. Wild-type KRAS is required for panitumumab efficacy in patients with metastatic colorectal cancer. J Clin Oncol. 2008 Apr 1;26(10):1626-34. doi: 10.1200/JCO.2007.14.7116. Epub 2008 Mar 3. PMID 18316791
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: FDA-approved Drug Labeling — http://www.vectibix.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 January 2004 through 16 March 2005. Data are up until the data cutoff of 15 March 2007.
Groups:
- Panitumumab Plus BSC: Panitumumab plus best supportive care (BSC). Panitumumab was administered by intravenous infusion at a dose of 6 mg/kg once every 2 weeks until participants developed progressive disease or were unable to tolerate study drug.
- BSC Alone: Best supportive care defined as the best care available as judged appropriate by the investigator and according to institutional guidelines, including antibiotics, analgesics, radiation therapy for pain control (limited to bone metastases), corticosteroids, transfusions, psychotherapy, growth factors, palliative surgery, or any symptomatic therapy as clinically indicated. For the purpose of this study, best supportive care does not include anti-neoplastic chemotherapy.
Period: Overall Study
Arm/Group | Panitumumab Plus BSC | BSC Alone
Started | 231 | 232
Received Study Drug | 229 | 0
Completed | 158 (Defined as participants who completed safety follow-up visit or who died.) | 206 (Defined as participants who completed safety follow-up visit or who died.)
Not Completed | 73 | 26
Not completed — Adverse Event | 5 | 2
Not completed — Disease Progression | 28 | 14
Not completed — Lost to Follow-up | 10 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Other | 27 | 6
Not completed — Non-compliance | 1 | 0
Not completed — Ongoing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panitumumab Plus BSC | BSC Alone | Total
Number analyzed (Participants) | 231 | 232 | 463
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.3) | 61.4 (10.8) | 61.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 84 | 169
  Male | 146 | 148 | 294
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 0 | 1 | 1
  Aborigine | 0 | 0 | 0
  Other | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White or Caucasian | 229 | 228 | 457
  Hispanic or Latino | 1 | 1 | 2
Region of Enrollment [Number; unit: participants] — Central and Eastern Europe includes the Czech Republic, Greece, Hungary, and the Slovak Republic. Rest of World includes Australia, Canada and New Zealand. Western Europe includes Austria, Belgium, France, Germany, Italy, Portugal, Spain, Switzerland, and the Netherlands.
  participants
    Central and Eastern Europe | 20 | 19 | 39
    Western Europe | 178 | 180 | 358
    Rest of World | 33 | 33 | 66
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 or 1 | 200 | 202 | 402
    2 | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Time
Description: Kaplan-Meier estimates of median time from randomization to either death or first observed disease progression, whichever occurred first. Participants were evaluated for tumor response according to modified Response Evaluation Criteria in Solid Tumors (RECIST) based on the response assessment from a blinded review of radiographic scans by the Independent Review Committee. Progressive disease defined as least a 20% increase in the sum of the longest diameters (SLD) of target lesions, taking as reference the nadir SLD recorded since the treatment started or the appearance of one or more new lesions, or the unequivocal progression of existing non-target lesions.
Time Frame: From randomization to the data cut-off date of 30 June 2005. The median follow-up time was 20.0 weeks in the panitumumab plus BSC group and 18.2 weeks in the BSC alone group.
Population: Intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 231 | 232
weeks | 8.0 [7.9 to 8.4] | 7.3 [7.1 to 7.7]
Statistical Analysis 1: Comparison: Panitumumab Plus BSC vs BSC Alone; Null hypothesis was no difference between treatment groups; Test type: Superiority or Other; p < 0.0001, Log Rank; Stratified by baseline IVRS ECOG performance status and geographic region

2. Secondary Outcome: Overall Survival
Description: Kaplan-Meier estimates of median time from randomization to death.
Time Frame: From randomization until the data cut-off date for overall survival of 15 March 2006. The median actual follow-up time was 30 weeks for the panitumumab plus BSC group and 31 weeks for the BSC alone group.
Population: Intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 231 | 232
months | 6.4 [6.1 to 7.7] | 6.3 [4.9 to 7.6]
Statistical Analysis 1: Comparison: Panitumumab Plus BSC vs BSC Alone; Null hypothesis was no difference between treatment groups; Test type: Superiority or Other; p = 0.806, Log Rank — This analysis was conducted contingent on a statistically significant difference in the primary outcome, and adjusted to an a priori threshold for statistical significance at a 4% level for a multiple comparison involving objective tumor response; Stratified by baseline IVRS ECOG performance status and geographic region

3. Secondary Outcome: Objective Tumor Response
Description: Defined as the number of participants with a confirmed complete or partial tumor response, confirmed by a scan no less than 4 weeks after the criteria for response were first met. Participants were evaluated for tumor response according to modified Response Evaluation Criteria in Solid Tumors (RECIST) based on the response assessment from a blinded review of radiographic scans by the Independent Review Committee. Complete Response (CR): Disappearance of all target and non-target lesions and no new lesions. Partial Response (PR): disappearance of all target lesions, and persistence of one or more non-target lesion(s) not qualifying for either CR or progressive disease, or, at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline SLD, with no progressive disease of non-target lesions.
Time Frame: From randomization until the data cutoff of 15 March 2007. The median follow-up time was 29.6 weeks in the panitumumab plus BSC group and 31.8 weeks in the BSC alone group.
Population: Intention-to-treat (ITT)
Measure: Number; unit: participants
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 231 | 232
participants | 22 | 0

4. Secondary Outcome: Duration of Response
Description: Kaplan-Meier estimate of the median time from first confirmed objective tumor response to first observed progression of disease or death due to progression of disease (whichever comes first).
Time Frame: as for outcome 3
Population: Intention-to-treat participants who had a confirmed objective tumor response. No objective tumor responses were observed in the BSC alone treatment arm.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 22 | 0
weeks | 18.4 [16.0 to 25.3] |

5. Secondary Outcome: Time to Response
Description: Time to response was defined as the time from randomization to first partial or complete response, subsequently confirmed ≥ 4 weeks after the criteria for response were first met.
Time Frame: as for outcome 3
Population: Intention-to-treat (ITT) participants who had a confirmed objective tumor response. No objective tumor responses were observed in the BSC alone treatment arm.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 22 | 0
weeks | 7.9 [7.3 to 10.6] |

6. Secondary Outcome: Time to Disease Progression
Description: Kaplan-Meier estimates of median time from randomization to disease progression or death due to disease progression (whichever occurs first)
Time Frame: as for outcome 3
Population: Intention-to-treat
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 231 | 232
weeks | 8.0 [7.9 to 8.9] | 7.3 [7.1 to 7.7]

7. Secondary Outcome: Time to Treatment Failure
Description: Kaplan-Meier estimate of the median time from randomization to the date the decision was made to end treatment for any reason.
Time Frame: as for outcome 3
Population: Intention-to-treat (ITT)
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 231 | 232
weeks | 9.0 [8.3 to 12.0] | 7.1 [6.4 to 7.6]

8. Secondary Outcome: Duration of Stable Disease
Description: Kaplan-Meier estimate of the median time from randomization to date of first observed progression of disease or death due to progression of disease (whichever comes first) for those participants with a best response of stable disease. Stable disease defined as neither sufficient shrinkage to qualify for a partial response nor sufficient increase to qualify for progressive disease taking as reference the nadir longest diameter since the treatment started, no unequivocal progression of existing non-target lesions, and no new lesions.
Time Frame: as for outcome 3
Population: Participants who had a best overall response of stable disease
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab Plus BSC | BSC Alone
Number analyzed (Participants) | 61 | 24
weeks | 24.0 [22.4 to 27.3] | 17.6 [15.4 to 25.6]

9. Post Hoc Outcome: Progression-free Survival Time (Wild-type KRAS)
Description: Kaplan-Meier estimates of median time from randomization to either death or first observed disease progression among participants with wild-type Kirsten Rat Sarcoma Virus Oncogene (KRAS) status. Participants were evaluated for tumor response according to modified Response Evaluation Criteria in Solid Tumors (RECIST) based on the response assessment from a blinded review of radiographic scans by the Independent Review Committee. Progressive disease defined as least a 20% increase in the sum of the longest diameters (SLD) of target lesions, taking as reference the nadir SLD recorded since the treatment started or the appearance of one or more new lesions, or the unequivocal progression of existing non-target lesions.
Time Frame: From randomization until the data cutoff of 15 March 2007. The median follow-up time in patients with wild-type KRAS was 36.8 weeks in the panitumumab plus BSC group and 35.7 weeks in the BSC alone group.
Population: Wild-type KRAS Efficacy Analysis Set, a subset of the Intention-to-Treat set with wild-type Kirsten Rat Sarcoma Virus Oncogene (KRAS) status.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Panitumumab Plus Best Supportive Care: Panitumumab plus best supportive care (BSC). Panitumumab was administered by intravenous infusion at a dose of 6 mg/kg once every 2 weeks until participants developed progressive disease or were unable to tolerate study drug.
Arm/Group | Panitumumab Plus Best Supportive Care | BSC Alone
Number analyzed (Participants) | 124 | 119
weeks | 12.3 [8.3 to 16.1] | 7.3 [7.0 to 7.7]

10. Post Hoc Outcome: Progression-free Survival Time (Mutant KRAS)
Description: Kaplan-Meier estimates of median time from randomization to either death or first observed disease progression among participants with mutant Kirsten Rat Sarcoma Virus Oncogene (KRAS) status. Participants were evaluated for tumor response according to modified Response Evaluation Criteria in Solid Tumors (RECIST) based on the response assessment from a blinded review of radiographic scans by the Independent Review Committee. Progressive disease defined as least a 20% increase in the sum of the longest diameters (SLD) of target lesions, taking as reference the nadir SLD recorded since the treatment started or the appearance of one or more new lesions, or the unequivocal progression of existing non-target lesions.
Time Frame: From randomization until the data cutoff of 15 March 2007. The median follow-up time in patients with mutant KRAS was 24.4 weeks in the panitumumab plus BSC group and 23.9 weeks in the BSC alone group.
Population: Mutant KRAS Efficacy Analysis Set, a subset of the Intention-to-Treat set with mutant Kirsten Rat Sarcoma Virus Oncogene (KRAS) status.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Panitumumab Plus Best Supportive Care | BSC Alone
Number analyzed (Participants) | 84 | 100
weeks | 7.4 [7.3 to 7.9] | 7.3 [6.3 to 7.9]

ADVERSE EVENTS:
Time Frame: First dose through maximum of safety FU or 30 days after last dose
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. Safety Analysis set includes all randomized patients, analyzed according to the treatment they actually received. Hence, 2 patients randomized to Panitumumab Plus BSC treatment group are analyzed in the BSC Alone group for safety.
Arm/Group | Panitumumab Plus BSC | BSC Alone
Serious Adverse Events (participants affected / at risk) | 101/229 | 62/234
Other Adverse Events (participants affected / at risk) | 224/229 | 171/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus BSC (N=229) | BSC Alone (N=234)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0
ENDOPHTHALMITIS (Eye disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 8 | 8
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 4 | 2
CONSTIPATION (Gastrointestinal disorders) | 7 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
DUODENAL STENOSIS (Gastrointestinal disorders) | 0 | 1
GASTRIC ULCER (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 11 | 4
MELAENA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 2
PERITONITIS (Gastrointestinal disorders) | 1 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 1
RECTAL DISCHARGE (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 1
VOMITING (Gastrointestinal disorders) | 4 | 5
ASTHENIA (General disorders) | 4 | 2
CATHETER RELATED COMPLICATION (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 14 | 6
HYPERTHERMIA (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0
OEDEMA (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PELVIC MASS (General disorders) | 1 | 0
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 1
PYREXIA (General disorders) | 1 | 8
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 0 | 2
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 5 | 4
HEPATOMEGALY (Hepatobiliary disorders) | 2 | 0
HEPATORENAL FAILURE (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 3 | 2
JAUNDICE (Hepatobiliary disorders) | 4 | 3
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
LIVER DISORDER (Hepatobiliary disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 1 | 0
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1 | 0
EYE INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 0
HAEMOPHILUS INFECTION (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 0 | 1
LUNG INFECTION (Infections and infestations) | 1 | 0
PARONYCHIA (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 2
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 0 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 2
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
ANOREXIA (Metabolism and nutrition disorders) | 3 | 1
CACHEXIA (Metabolism and nutrition disorders) | 2 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 9
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 | 24
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO PLEURA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO SPINE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PERITONEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR INVASION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
TUMOUR NECROSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0
COMA (Nervous system disorders) | 2 | 0
COMA HEPATIC (Nervous system disorders) | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 2 | 0
EPILEPSY (Nervous system disorders) | 2 | 0
HEMIPARESIS (Nervous system disorders) | 2 | 1
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 2 | 2
LETHARGY (Nervous system disorders) | 1 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
SOMNOLENCE (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 | 1
STUPOR (Nervous system disorders) | 0 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
ALCOHOLISM (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 2
DEPRESSION (Psychiatric disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0
OLIGURIA (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 1 | 0
FEMALE GENITAL TRACT FISTULA (Reproductive system and breast disorders) | 0 | 1
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 1
PERINEAL PAIN (Reproductive system and breast disorders) | 0 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0
AXILLARY VEIN THROMBOSIS (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 0
HAEMORRHAGE (Vascular disorders) | 1 | 0
JUGULAR VEIN THROMBOSIS (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panitumumab Plus BSC (N=229) | BSC Alone (N=234)
ANAEMIA (Blood and lymphatic system disorders) | 12 | 6
GROWTH OF EYELASHES (Eye disorders) | 13 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 56 | 36
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 19 | 16
CONSTIPATION (Gastrointestinal disorders) | 43 | 21
DIARRHOEA (Gastrointestinal disorders) | 48 | 26
NAUSEA (Gastrointestinal disorders) | 51 | 35
STOMATITIS (Gastrointestinal disorders) | 15 | 2
VOMITING (Gastrointestinal disorders) | 41 | 27
ASTHENIA (General disorders) | 28 | 25
FATIGUE (General disorders) | 59 | 34
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 13 | 3
MUCOSAL INFLAMMATION (General disorders) | 14 | 2
OEDEMA PERIPHERAL (General disorders) | 27 | 13
PYREXIA (General disorders) | 37 | 24
HEPATOMEGALY (Hepatobiliary disorders) | 12 | 8
JAUNDICE (Hepatobiliary disorders) | 13 | 7
PARONYCHIA (Infections and infestations) | 57 | 0
WEIGHT DECREASED (Investigations) | 12 | 3
ANOREXIA (Metabolism and nutrition disorders) | 63 | 44
BACK PAIN (Musculoskeletal and connective tissue disorders) | 24 | 16
ANXIETY (Psychiatric disorders) | 14 | 7
INSOMNIA (Psychiatric disorders) | 15 | 14
COUGH (Respiratory, thoracic and mediastinal disorders) | 34 | 17
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 36 | 28
ACNE (Skin and subcutaneous tissue disorders) | 31 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 131 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 23 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 150 | 2
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 41 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 22 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 132 | 4
RASH (Skin and subcutaneous tissue disorders) | 51 | 2
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 21 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 45 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 13 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.